CLINICAL TRIAL: NCT04748133
Title: Acupuncture for Enhancing Recovery and Attenuating Postoperative Nausea and Vomiting After Middle Ear Surgeries: A Randomized Controlled Trial
Brief Title: Acupuncture for Recovery and Postoperative Nausea and Vomiting After Middle Ear Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mahmoud Abd Allah Zakzouk, Lecturer of Anesthesia & Surgical Intensive Care, Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6658
Record Dates: First submitted 2021-02-08; First posted 2021-02-10 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Treatment Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture (Active Comparator): Patients in the acupuncture group will receive a standardised treatment with 12 needles (sharp tip, stainless steel needles, size 0.3 X 40 mm) at 7 acupuncture points Du 26 and Ren 17 (on the middle body line), and bilateral LI 4, HE 7, LV 3, ST 36 and PC 6). Application of the needles is performed by a licensed medical acupuncturist.
  The needles will be inserted after endotracheal intubation and mechanical ventilation and will be removed immediately before patient extubation.
  Interventions: Device: acupuncture needles
- placebo (Placebo Comparator): no treatment
  Interventions: Other: placebo

INTERVENTIONS:
Device: acupuncture needles — Site of acupuncture points:
  * Du 26: At junction of the upper and middle third of philtrum.
  * Ren 17: On the midline level with the 4th intercostal space midway between the nipples.
  * LI4 (Large Intestine 4): On the dorsum of the hand, between the 1st and 2nd metacarpal bones
  * HT7 (Heart 7): On the ulnar end of the transverse crease of the wrist, in the small depression between the pisiform and ulna bones
  * LV3 (Liver 3): On dorsum of the foot in a depression distal to the junction of the 1st and 2nd metatarsal bones.
  * ST36 (Stomach 36): Antero-lateral leg, 1 middle-finger breadth next to the anterior crest of tibia, 3 cun under the depression lateral to the patellar ligament.
  * PC6 (Pericardium 6): Palmar aspect of the forearm, between the tendons, 2 cun away from the transverse crease of the wrist
  Arms: acupuncture
Other: placebo — no treatment
  Arms: placebo

SUMMARY:
Modern surgery management needs increasing operating room turnover and more ambulatory surgery. In order to come over this challenge, the recovery needs to be optimized. Enhancing recovery could be achieved by preventing postoperative pain and postoperative nausea and vomiting. Middle ear surgery is a common ambulatory surgery with increasing occurrence of postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Sample size: as percent of vomiting following acupuncture and following standard anesthesia is 0.13% and 29.2% respectively so sample size is 58 (29 in each group). Sample is calculated using open epi program with confidence level 95% and power 80%.

Patients in Group C (control group) (n=29): will receive no treatment. While patients in Group A (Acupuncture group) (n=29): will receive needle acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Age: 21-60 years old.
* Sex: both sex (males or females).
* Physical status: ASA 1& II.
* BMI = (20-30 kg/m2).
* Type of operations: elective unilateral middle ear surgeries such as tempanoplasty, stapedectomy and mastedictomy.

Exclusion Criteria:

* Altered mental state
* Patients with Drug abuse or alcohol.
* Patients with on antipsychotic drugs, regular antiemetic therapy or receiving antiemetic 24 hour before surgery.
* Patients with pre-treatment with acupuncture or trigger point injection.
* Pregnancy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative nausea and vomiting | up to 24 hours postoperative
  Postoperative nausea and vomiting impact scale score . Questions Answers score Did you have vomiting or dry retching? No 0 Once 1 Twice 2 Three or more times 3
  Have you experienced a feeling of nausea? If yes, has it interfered with your daily activities? Not at all 0 Sometimes 1 Often/most of the times 2 All the time 3
  Summation of numerical answer to question 1 plus 2 equal the PONV impact scale. PONV Impact Scale Score of ≥5 represents clinically important PONV

SECONDARY OUTCOMES:
extubation time | up to 10 minutes postoperative
  time from discontinuation of isoflurane to extubation
recovery time | up to 30 minutes postoperative
  time from discontinuation of isoflurane to first response to verbal command
The time of discharge | up to 30 minutes postoperative
  The time from arrival to PACU to discharge to the ward) according to Modified Aldert score Modified Aldert score . Assessment item Condition Grade Activity, able to move, voluntarily or on command 4 extremities 2 2 extremities 1 No 0
  Breathing Able to breathe deeply & cough freely 2 Dyspnea, shallow or limited breathing 1 Apnea 0 Consciousness Fully awake 2 Arousable on calling 1 Unresponsive 0
  Circulation (blood pressure) ±20% of pre-anesthesia level 2
  * 20% to 49% of pre-anesthesia level 1
  * 50% of pre-anesthesia level 0 SPO2 Maintain SPO2 >92% in ambient air 2 Maintain SPO2 >90% with O2 1 Maintain SPO2 <90% with O2 0
  Patient having a score of 9 or higher is discharged
The total number of rescue antiemetic (metoclopramide) | in the first 24 hour postoperative
  Any patient will receive 10 mg intravenous metoclopramide immediately if there is nausea and vomiting
Postoperative Pain | up to 30 minutes, 2 hours and 4 hours postoperative
  Visual Analogue Scale (VAS) . A commonly used scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border. The patient is instructed to make a mark along the line to represent the intensity of pain currently being experienced. IV paracetamol 1 gm every 6hs as a protocol for pain management and IV pethidine 30 mg as rescue analgesic will be given if VAS ≥ 4. Total doses and number of analgesics will be recorded
number of participant with side effects of acupuncture | up to 24 hours postoperative
  bleeding, soreness, or bruising at the site of needle insertion

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Zakzouk, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt